CLINICAL TRIAL: NCT03034330
Title: A Two-Tier Care Management Program to Empower Stroke Caregivers in Hong Kong: A Randomized Controlled Trial
Brief Title: A Two-Tier Care Management Program to Empower Stroke Caregivers in Hong Kong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Vivian W.Q. Lou, Director, Sau Po Center on Ageing, Faculty of Social Science, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UW16-1019
Record Dates: First submitted 2017-01-13; First posted 2017-01-27 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Stroke
Keywords: informal care; empowerment; family-focused intervention; stroke rehabilitation
MeSH Terms: conditions — Stroke; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Two-Tier Stroke Family Empowerment (Experimental): The intervention is individualized, tailor-made according to caregivers' needs. The intervention will last for 2 to 3 months with 6 to 10 weekly sessions at the home of caregivers or stroke survivors. Each session will last for 60 to 90 minutes. The care managers will determine the intensity of the intervention after the initial family assessment.
  Interventions: Other: Two-Tier Stroke Family Empowerment
- Volunteer Support Psychoeducation (Active Comparator): The intervention will last for 2 months with 4 weekly sessions at the home of caregivers or stroke survivors in the first month and 2 telephone contacts in the second month (6 contact points in total). Each session will last for 60 to 90 minutes. Care managers will not provide any direct intervention for participants in the control group.
  Interventions: Other: Volunteer Support Psychoeducation

INTERVENTIONS:
Other: Two-Tier Stroke Family Empowerment — The family-based care management intervention will be implemented in two tiers. The first tier is the Family Care Management that a care manager is responsible for empowering family caregivers to support their stroke survivors through reorganizing family roles, enhancing family functioning, and maximizing their family and community resources. The second tier is led by trained volunteers who are responsible for increasing the capacity of caregivers for the mastery of stroke care by providing psychoeducation, skill-training, and social support. Each caregiver participant will be assigned a care manager and a volunteer. All care managers who are social workers from the participating centres have undergone 4-day training to improve their knowledge of stroke and skills required for the intervention. Similarly, volunteers have undergone 6.5-day training to equip them with the knowledge and skills to conduct the intervention.
  Arms: Two-Tier Stroke Family Empowerment
Other: Volunteer Support Psychoeducation — The active control group will receive a standard, non-family-based psychoeducation intervention provided by the trained volunteers under the supervision of care managers. It will provide 4 in-home visits and 2 telephone follow-up interviews about psychoeducation for caregivers of stroke survivors.
  Arms: Volunteer Support Psychoeducation

SUMMARY:
This study intends to develop a family-based care management intervention with primary aims to provide time-limited support for family caregivers affected by stroke and to empower caregivers through enhancing the family adaptation and functioning and increasing their capacity of stroke care. The objectives include:

1. To examine the effectiveness of the proposed family-based intervention to improve family, caregiver, and service outcome.
2. To examine the cost-effectiveness of the proposed family intervention.

It is hypothesized that comparing to the control group, the experimental group participants will have more and significant outcome.

DETAILED DESCRIPTION:
This study will recruit 300 caregivers of first stroke survivors to involve in the intervention and employ a randomized controlled trial (RCT) to assign the caregivers into the intervention group and active control group. Each group will have 150 caregivers. The intervention is individualized, tailor-made according to caregivers' needs. Care managers will conduct an initial family need assessment with caregivers to determine their care plan. The intervention will last for 2 to 3 months with 6 to 10 weekly sessions. If the caregiver participants' family member with stroke (stroke survivors) agrees to and is competent enough( see Eligibility Criteria Criteria), they will also be invited to take part in up to 4 intervention sessions.

The active control group will receive a standard, non-family-based psychoeducation intervention provided by the trained volunteers under the supervision of care managers. The active control group will not involve stroke survivors. Therefore, a maximum of 150 stroke survivors will be involved in the intervention.

Both caregivers participants (300) and their family members with stroke (300) will be asked to do questionnaires before (T1), immediately after (T2) and 2 months after (T3) the intervention. The intervention and the questionnaire interview will take place at the homes of participants.

The participation of the stroke survivors in the intervention and the questionnaire interview will not affect the involvement of their caregivers in this study. In other words, caregivers can still take part in the intervention and the questionnaire interview if their family members with stroke refuse to or are not competent ( see Eligibility Criteria Criteria) to take part in this study.

No drug usage and medical treatment will be involved in the study. Intervention and questionnaires do not impose any physical or medical risk to participants. The only possible problem may be caregivers may feel a little tired after the intervention. Participants can voluntarily drop out the study at any time, without giving any reason, without my medical care or original rights being affected.

Both the effectiveness and the cost-effectiveness will be evaluated in this study (See Outcome Measures). Chi-square or independent t-tests will be used to examine the differences in the baseline characteristics between the intervention and control groups. To assess the effectiveness of the intervention, regression analysis will be used to compare the difference in outcomes between the intervention and control groups, controlling for the effect of potential covariates. Recruitment rate, drop-out rate and missing data will also be examined and reported.

The principal investigator will be responsible for keeping of the personal data during and after the study. The data will be for academic and clinical research only and will be kept for up to 5 years and will be destroyed after that.

ELIGIBILITY:
Inclusion Criteria:

* A stroke caregiver is eligible to participate in the study if:

  1. He / She is a Chinese adult aged 18 or above;
  2. He / She has a family member has the first stroke (ischaemic or haemorrhagic stroke) at the age of 50 or above and has been discharged from the acute hospital for no more than 6 months;
  3. He / She provides care or being with the stroke survivor for no less than two hours per day after discharge from the acute hospital;
  4. He / She reports significant caregiver burden as measured by the 12-item Zarit Burden Interview (a total score ≥ 12).

A stroke survivor is eligible to participate in the study if:

1. He / She is a Chinese adult aged 50 or above;
2. He / She has been discharged from the acute hospital for no more than 6 months;
3. His / Her family caregiver participates in this study;
4. He/ She is able to communicate with interventionists and interviewers;
5. He/ She is competent to give written informed consent.

Stroke survivors whose caregivers in the intervention group will receive both the intervention and the questionnaire interviews. Stroke survivors whose caregiver in the control group will only need to take part in the questionnaire interview.

Exclusion Criteria:

* A stroke caregiver will be excluded from participation if:

  1. His / Her family member has a transient ischaemic attack without a major ischaemic or haemorrhagic stroke;
  2. His / Her family member with stroke is residing in a residential care facility after discharge from the acute hospital;
  3. He / She is diagnosed as having Alzheimer's disease or other dementias;
  4. He / She is unable to understand Cantonese.

A stroke survivor is not eligible to participate in the study if:

1. He / She is residing in a residential care facility after discharge from the acute hospital;
2. He/ She has a transient ischaemic attack without a major ischaemic or haemorrhagic stroke;
3. His / Her family caregiver refuses to participate in this study;
4. He/ She is not able to communicate with interventionists and interviewers;
5. He/ She is not competent to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2017-01; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Family Role Performance measured by the Family Role Performance Scale (Questionnaire) | 6 months
  Family Role Performance Scale: The research team develops this scale to measure the frequency and ability of the family member to perform six major family roles, which are advisor, emotional connector, breadwinner, caretaker, decision maker and caregiver. The scale has two parts. The first part contains 6 items and asks participants how often they perform the six family roles. The second part contains 6 items and asks participants to rate their performance regarding to the family roles.
Care Management Strategies measured by the Care Management Strategies Scale (Questionnaire) | 6 months
  Care Management Strategies Scale: This is a 5-point Likert scale developed by the research team to find out the care management behaviors proposed by stroke caregivers. The scale contains 18 items.
Family Caregiver Conflict measured by Family Caregiver Conflict Scale (FCCS) (Questionnaire) | 6 months
  Family Caregiver Conflict Scale (FCCS): This is a 5-Likert-type scale with 15 items to assess family conflict due to stroke. It has four subscales: communication, problem solving, general family functioning, and perceived criticism (Clark, Shields, Aycock, & Wolf, 2003).
Family Function measured by the Family Assessment Device-General Functioning Scale (FAD-GF) (Questionnaire) | 6 months
  Family Assessment Device-General Functioning Scale (FAD-GF): This study will use the 12-item general functioning of the McMaster Family Assessment Device (Epstein, Baldwin, & Bishop, 1983) to measure the family functioning of caregivers. Responses are given using a 4-point Likert scale (1 = strongly agree to 4 = strongly disagree).

SECONDARY OUTCOMES:
Caregiver Burden measuewd by the Cantonese Short Version of Zarit Burden Interview (questionnaire) | 6 months
  Cantonese Short Version of Zarit Burden Interview: It is a spoken Cantonese version of the 12-item Zarit Burden Interview (ZBI) to assess the burden of Chinese dementia caregivers in clinical and social care settings (Tang et al., 2015). Participants answer on a 5-point scale ranging from 0 (never) to 4 (very frequently) regarding how often they feel burdened by their caregiving duties (e.g., "feel stressed between caregiving and meeting other responsibilities").
Depressive symptoms measured by the The Patient Health Questionnaire-9 (PHQ-9) (Questionnaire) | 6 months
  The Patient Health Questionnaire-9 (PHQ-9): The PHQ-9 is a reliable and valid instrument for assessing depressive symptoms of the general population in Hong Kong. It has 9 questions and was developed to correspond to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, criteria for major depression (Yu, Tam, Wong, Lam, & Stewart, 2012).
Ambivalence between caregivers and care receivers measured by the Caregiving Ambivalence Scale (Questionnaire) | 6 months
  Caregiving Ambivalence Scale: This scale is based on the Intergenerational Ambivalence Scale (Guo, Chi, & Silverstein, 2013) to measure the level of ambivalence between caregivers and care receivers. The scale for caregivers has six items, three asking the positive components and three asking the negative components of their relationships (0 = not at all, 1 = somewhat, and 2 = very). The scale for care receivers has one more item than the caregiver scale asking the question "Do you have tense and strained feelings when think about your relationship with your domestic help?"
The mental or affective state of caregivers in relation to stressful caregiving experience measured by the Positive Aspects of Caregiving (PAC) (Questionnaire) | 6 months
  Positive Aspects of Caregiving (PAC): PAC scale measures the mental or affective state of caregivers in relation to stressful caregiving experience (Tarlow et al., 2004). The scale contains 11 questions and responses are given using a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree) (Lou, Lau, & Cheung, 2015).
Social network of caregivers measured by the Lubben Social Network Scale (LSNS) (Questionnaire) | 6 months
  Lubben Social Network Scale (LSNS): The original Chinese versions of the Lubben Social Network Scale (LSNS) comprises 10 questions that rate the level of social support. Each question ranges from 0 to 5; higher scores indicate a better social network (Lubben, 1988).
Contemporary filial piety of caregivers measured by the Contemporary Filial Piety Scale (CFPS-10) (Questionnaire) | 6 months
  Contemporary Filial Piety Scale (CFPS-10): This is a 5-point Likert scale scale with 10-items to assess contemporary filial piety in the 21st century. It tests two factors. The first factor, Pragmatic Obligations, contained 6 filial behavior items related to practical and pragmatic caregiving. The second factor, Compassionate Reverence, contained 4 filial attitude items related to emotional caregiving (Lum et al., 2015).
Stroke knowledge of caregivers measured by the Stroke Knowledge Test (SKT) (Questionnaire) | 6 months
  Stroke Knowledge Test (SKT): The stroke health literacy of caregivers is measured by a Stroke Knowledge Test (SKT) tailored for this project by a physician with expertise in neurology who is in charge of a stroke clinic in a major public hospital in Hong Kong. The Test has 9 questions.
Self-rated Health measured by a question to rate their health (Questionnaire) | 6 months
  Self-rated Health: One question will be asked for caregivers and stroke survivors to rate their health "General speaking, what do you think about your physical health?"
Health-related quality of life measured by SF-12 Health Survey (SF-12) (Questionnaire) | 6 months
  SF-12 Health Survey (SF-12): This is a valid and widely used scale with 12 items to measure the health-related quality of life (HRQOL) among the general Chinese population in Hong Kong (Lam, Wong, Lam, Lo, & Huang, 2010).
Degree of disability or dependence in the daily activities of people who have suffered from a stroke measured by the Simplified Modified Rankin Scale (Questionnaire) | 6 months
  Simplified Modified Rankin Scale: Modified Rankin Scale is a commonly used and reliable scale for measuring the degree of disability or dependence in the daily activities of people who have suffered from a stroke. The simplified version preserves the original construct and validity of the Modified Rankin Scale and makes it relatively simple and short with only 5 questions. The simplified version has good reliability (Bruno, et al., 2011).
The rate of inpatient hospital admission of stroke survivors | 6 months
Number of specialist outpatient received by stroke survivors | 6 months
Number of accident and emergency service received by stroke survivors | 6 months
Number of medicines received by stroke survivors | 6 months
Number of hospital rehabilitation service received by stroke survivors | 6 months
Number of home care service received by stroke survivors | 6 months
  Social care services include home care service, day care service, community rehabilitation service, residential care service (admission after study intake).
Number of day care service received by stroke survivors | 6 months
Number of community rehabilitation service received by stroke survivors | 6 months
Number of residential care service received by stroke survivors(admission after study intake) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lou Vivian, Vivian, Principal Investigator — Sau Po Center on Ageing, HKU
Locations (1):
- Sau Po Center on Ageing HKU, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data collected in this study will be published and submitted to academic journals to share with other researchers.

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082
- [Derived] Lou VW, Tang JYM, Lau GKK, Lum TYS, Fong K, Ko RWT, Cheng CYM, Fu JY, Chow ESL, Chu ACK, Hui E, Ng WWL, Chan FHW, Luk CC, Kwok TK. Effectiveness of a Two-Tier Family-Oriented Intervention in Enhancing the Family Functioning and Care Capacity of the Family Caregivers of Stroke Survivors: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 May 28;10(5):e16703. doi: 10.2196/16703. PMID 34047707